CLINICAL TRIAL: NCT04113096
Title: Use of Dibenzyl Trisulphide as a Chemotherapeutic Agent in Stage Four Cancer of the Breast, Prostate, Cervix and Colon
Brief Title: Dibenzyl Trisulphide (GUINEAHEN WEED) for Stage IV Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of The West Indies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ECP 250 - 15/16
Record Dates: First submitted 2018-11-26; First posted 2019-10-02 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2018-10

CONDITIONS: Stage IV Prostate Cancer; Stage IV Colon Cancer; Stage IV Breast Cancer; Stage IV Cancer of the Cervix
MeSH Terms: conditions — Prostatic Neoplasms; Colonic Neoplasms; Breast Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: For each condition there will be two arms of treatment. One arm will receive the investigational product and standard of care the other arm will receive placebo and standard of care
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Breast Cancer Stage IV (Experimental): Stage IV Breast Cancer: Dibenzyl trisulphide capsules (20mg once daily)/6 months
  Interventions: Drug: Dibenzyl trisulphide capsules; Drug: Stage IV Breast Cancer Placebo
- Colon Cancer Stage IV (Experimental): Stage IV Colon Cancer:Dibenzyl trisulphide capsules (20 mg one daily for 6 months
  Interventions: Drug: Dibenzyl trisulphide capsules; Drug: Stage IV: Colon Cancer Placebo
- Cervical Cancer Stage IV (Experimental): Stage IV Cancer of the Cervix: Dibenzyl trisulphide capsules (20 mg once daily) for 6 months
  Interventions: Drug: Dibenzyl trisulphide capsules; Drug: Cervical Cancer Stage IV Placebo
- Cancer of the Prostate Stage IV (Experimental): Stage IV Prostate cancer:Dibenzyl trisulphide capsules (20 mg once daily) for 6 months
  Interventions: Drug: Dibenzyl trisulphide capsules; Drug: Cancer of the Prostate Placebo

INTERVENTIONS:
Drug: Dibenzyl trisulphide capsules — 20 mg once daily for 6 months
  Other Names: Guineahen Weed capsules
  Arms: Breast Cancer Stage IV
Drug: Dibenzyl trisulphide capsules — 20 mg once daily for 6 months
  Other Names: Guineahen Weed capsules
  Arms: Colon Cancer Stage IV
Drug: Dibenzyl trisulphide capsules — 20 mg once daily for 6 months
  Other Names: Guineahen Weed capsules
  Arms: Cervical Cancer Stage IV
Drug: Dibenzyl trisulphide capsules — 20 mg once daily for 6 months
  Other Names: Guineahen Weed capsules
  Arms: Cancer of the Prostate Stage IV
Drug: Stage IV Breast Cancer Placebo — 20 mg once daily for 6 months
  Other Names: Placebo
  Arms: Breast Cancer Stage IV
Drug: Stage IV: Colon Cancer Placebo — 20 mg once daily for 6 months
  Other Names: Placebo
  Arms: Colon Cancer Stage IV
Drug: Cervical Cancer Stage IV Placebo — 20 mg once daily for 6 months
  Other Names: Placebo
  Arms: Cervical Cancer Stage IV
Drug: Cancer of the Prostate Placebo — 20 mg once daily for 6 months
  Other Names: Placebo
  Arms: Cancer of the Prostate Stage IV

SUMMARY:
This study is being done to find the effect of Dibenzyl Trisulphide (active ingredient in Guinea Hen Weed in combination in patients with stage four cancer of the breast, prostate, cervix and colon.

DETAILED DESCRIPTION:
There have been many claims of the value of Guinea Hen weed in the treatment of different cancers. The preparation is readily available and used locally. The team proposes to validate the studies done on cancer cell lines by conducting a clinical trial to determine the clinical benefit in advanced and metastatic cancers.

ELIGIBILITY:
Inclusion Criteria:

* Age: Greater than 12 years.
* Documented histologic evidence of cancer
* Staged as stage IV
* World Health Organization (WHO) Performance Status of between 0 and 2
* Radiological confirmation of metastases with bone scan or X ray, CT and/or MRI scan Exclusion Criteria

  * Cancer stages less than stage 4
  * Pregnant women
  * Children 0 - 12 years

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Prostate Cancer | Every 8 weeks up to 52 weeks
  50% change in the Prostate Specific Antigen Response (PSA)
Breast Cancer | Every 8 weeks up to 52 weeks
  Changes in size of the metastatic legions
Colon Cancer | Every 8 weeks up to 52 weeks
  50% change in the Carcinoembryonic Antigen (CEA)
Cervical Cancer | Every 8 weeks up to 52 weeks
  50% change in renal function (Renal output)

SECONDARY OUTCOMES:
Haemoglobin Red Cell Test | Every 8 weeks upto 52 weeks
  Blood - haemoglobin red cell count grams/decilitre
Blood Platelets Tests | Every 8 weeks upto 52 weeks
  Blood; platelet count per microlitre
Blood urea Tests | Every 8 weeks upto 52 weeks
  Blood Urea Nitrogen
Blood Creatinine | Every 8 weeks upto 52 weeks
  Amount of creatinine in the blood
Blood Electrolytes | Every 8 weeks upto 52 weeks
  Amount of electrolytes in the blood
Blood Calcium | Every 8 weeks upto 52 weeks
  Amount of calcium in the blood
Blood Phosphorus | Every 8 weeks upto 52 weeks
  Amount of phosphorus in the blood
Prothrombin Test | Every 8 weeks upto 52 weeks
  Blood prothrombin time (PT).
Partial Prothrombin Test | Every 8 weeks upto 52 weeks
  Partial thromboplastin time( PTT).
White Blood Cell Test | every 8 weeks up to 52 weeks
  white cell count per microlitre
Computed Tomography (CT) Scan | Every 8 weeks up to 52 weeks
  A pelvis baseline scan and level of metastases quantified by a single radiologist.
Nuclear bone scintigraphy | every 8 weeks up to 52 weeks
  A bone scintigraphy or X-ray to show number and site of metastases noted
Bilirubin Direct test | Every 8 weeks up to 52 weeks
  Bilirubin direct, mmol per litre
Bilirubin Indirect test | Every 8 weeks up to 52 weeks
  Bilirubin indirect mmol per litre
Alkaline Phosphate level test (ALP) | Every 8 weeks up to 52 weeks
  Amount of Alkaline Phosphate enzyme in blood units per litre
Aspartate Aminotransferase test | Every 8 weeks up to 52 weeks
  Level of the aspartate aminotransferase enzymes in the blood units per litre
Gamma-glutamyl transferase test | Every 8 weeks up to 52 weeks
  Level of the Gamma-glutamyl transferase units per litre
Lactate dehydrogenase test | Every 8 weeks up to 52 weeks
  Level of Lactate dehydrogenase units per litre
Respiration | Every 8 weeks up to 52 weeks
  Number of breaths per minute
Temperature measurement | Every 8 weeks up to 52 weeks
  Temperature; degrees centigrade
Pulse | Every 8 weeks up to 52 weeks
  Pulse-beats per minute
Cancer Survival Curves | Every 8 weeks up to 52 weeks
  Proportion of patients alive after administration of intervention

CONTACTS AND LOCATIONS:
Overall Officials: LAD Williams, Principal Investigator — University of the West Indies, Mona
Locations (1):
- Faculty of Medial Sciences, Kingston, Jamaica